CLINICAL TRIAL: NCT03731390
Title: A Phase I Clinical Study for Evaluating the Safety, Pharmacokinetics, and Preliminary Efficacy of Repeated Doses, Dose Escalation of GR1405 Injection in Patients With Advanced Solid Tumor or Lymphoma
Brief Title: GR1405 Injection in Patients With Advanced Solid Tumor or Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shi Yuankai, Vice-president, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GR1405-002
Record Dates: First submitted 2018-11-02; First posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Tumor, Solid; Lymphoma
Keywords: programmed death ligand-1 (PD-L1)
MeSH Terms: conditions — Neoplasms; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GR1405 injection 3 mg/kg (Experimental): According to the patient's weight, the dose of this group is 3mg/kg.
  Interventions: Drug: GR1405 injection
- GR1405 injection 10 mg/kg (Experimental): According to the patient's weight, the dose of this group is 10mg/kg.
  Interventions: Drug: GR1405 injection
- GR1405 injection 20 mg/kg (Experimental): According to the patient's weight, the dose of this group is 20mg/kg.
  Interventions: Drug: GR1405 injection
- GR1405 injection 30 mg/kg (Experimental): According to the patient's weight, the dose of this group is 30mg/kg.
  Interventions: Drug: GR1405 injection

INTERVENTIONS:
Drug: GR1405 injection — Intravenous administration according to the patient's weight. All dose groups were administered once every 2 weeks.
  Other Names: PD-L1 monoclonal antibody

SUMMARY:
This is a Phase I clinical study for evaluating the safety, pharmacokinetics, and preliminary efficacy of repeated doses, dose escalation of GR1405 injection in patients with advanced solid tumor or lymphoma

DETAILED DESCRIPTION:
To evaluate the tolerability, safety, pharmacokinetics, and preliminary efficacy of GR1405 injection monotherapy in an open, non-controlled, escalating trial design in patients with advanced solid tumors or lymphomas. Four dose levels (3 mg/kg, 10 mg/kg, 20 mg/kg, and 30 mg/kg) were evaluated at this stage.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with local advanced, recurrent or metastatic solid tumors confirmed by cytology or histology Lymphoma patients with pathological confirmation, and the above pat reients failed to standard treatment failure or had no standard treatment;
2. Aged 18 to 75 years men and women;
3. At least one measurable or evaluable lesion according to Response Evaluation Criteria in Solid Tumors v1.1(RECIST v1.1 )(solid tumor) or Lugano 2014 criteria (lymphoma);
4. Eastern Cooperative Oncology Group(ECOG)≤ 1
5. Female or male subjects of reproductive age and their mate are willing to take effective contraceptive measures for the entire treatment period and 6 months after the treatment;
6. With sufficient organ and bone marrow function;
7. At least 4 weeks after the last anti-tumor treatment before the first administration;
8. The patient or his legal representative signs a written informed consent.

Exclusion Criteria:

1. Have experienced any National Cancer Institute Common Terminology Criteria for Adverse events (NCI CTCAE) v4.03 or greater than 3 grade irAE during previous immunotherapy treatment;
2. Has received any anti-PD-1(programmed death 1) or anti-PD-L1 antibody treatment;
3. Subjects with other malignant tumors previously or concurrently ;
4. Female patients with pregnancy or lactation;
5. Women/men who have fertility refusal to adopt contraception during the trial period;
6. Subjects with serious disease or complications, such as gastrointestinal bleeding, intestinal obstruction, intestinal paralysis, interstitial pneumonia, pulmonary fibrosis, renal failure, glaucoma, uncontrolled diabetes (CTCAE= 4.03: fasting blood glucose level ≥ 2), and with active infection;
7. Had history of acute myocardial infarction, unstable angina pectoris, stroke or transient ischemic attack 6 months before the screening ,grade 2 or above congestive heart failure devised by the New York Heart Association (NYHA);
8. Subjects with symptomatic brain metastases or mental disorders;
9. Subjects with abnormal levels of serum calcium, magnesium, potassium and have clinical significance;
10. Subjects with history of immunodeficiency, including human immunodeficiency virus(HIV)-positive, suffering from other acquired, congenital immunodeficiency disease, or history of organ transplantation;
11. Subjects with active hepatitis B (HBsAg and/or HBcAb positive, and HBV DNA titer in peripheral blood was greater than 1 x 103 IU/ml), and/or hepatitis C;
12. Subjects who have alcohol addiction and/or drug abuse;
13. Subjects with bleeding or coagulation dysfunction in the past 3 months (Prothrombin time(PT)>1.5×upper limit of normal(ULN); activated partial thromboplastin time(APTT)>1.5×ULN; thrombin time(TT)>1.5×ULN);
14. Subjects with allergic constitution or allergic to known components of the drug;
15. Those who received other clinical trial drug therapy within 1 month before the first administration;
16. Receive a live attenuated vaccine within 4 weeks prior to the first dose of study treatment or during the study period;
17. Other subjects judged by the investigator to be ineligible for enrollment in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 2 weeks
  Maximum tolerated dose of GR1405 injection
Adverse Events | Approximately 3 years
  Number of Participants With Treatment-Emergent Adverse Events as Assessed by CTCAE v4.03

SECONDARY OUTCOMES:
maximum concentration (Cmax) | Approximately 2 years
  the maximum exposure to a biologically active physica
Duration of response (DOR) | Approximately 3 years
  DOR by RECIST v. 1.1 or Lugano 2014, the time between the initial response to therapy and subsequent disease progression or relapse
Objective Response Rate(ORR) | Approximately 3 years
  Objective Response Rate(ORR) by RECIST v. 1.1 or Lugano 2014, ORR=complete response(CR) + partial response(PR)
Progression free survival(PFS) | Approximately 3 years
  Progression free survival(PFS) by RECIST v. 1.1 or Lugano 2014, a patient lives with the disease but it does not get worse. In a clinical trial, measuring the progression-free survival is one way to see how well a new treatment works
Immunogenicity | Approximately 3 years
  the ability to elicit an immune response of GR1405 injection,
Recommended dose for Phase II trial(RP2D) | Approximately 3 years
  The MTD is one dose level below the lowest dose tested in which 2 or more patients experienced dose-limiting toxicity(DLT) attributable to the study drug. The MTD will be the RP2D
AUC0-t | Approximately 2 years
  Area under the curve in the period from 0 to t
AUC0-∞ | Approximately 2 years
  Area under the curve in the period from 0 to ∞
AUCss | Approximately 2 years
  Area under the curve of Steady-State Plasma Concentrations
T max | Approximately 2 years
  the time of occurrence of peak drug concentration
t 1/2 | Approximately 2 years
  the time of half-life of the drug
apparent volume of distribution (Vz) | Approximately 2 years
  the volume of fluid that would be required to contain the amount of drug in the body
clearance(CL) | Approximately 2 years
  the rate of elimination of the drug in vivo

CONTACTS AND LOCATIONS:
Overall Officials: yuankai Shi, M.D., Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute/Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Khoueiry AB, Sangro B, Yau T, Crocenzi TS, Kudo M, Hsu C, Kim TY, Choo SP, Trojan J, Welling TH Rd, Meyer T, Kang YK, Yeo W, Chopra A, Anderson J, Dela Cruz C, Lang L, Neely J, Tang H, Dastani HB, Melero I. Nivolumab in patients with advanced hepatocellular carcinoma (CheckMate 040): an open-label, non-comparative, phase 1/2 dose escalation and expansion trial. Lancet. 2017 Jun 24;389(10088):2492-2502. doi: 10.1016/S0140-6736(17)31046-2. Epub 2017 Apr 20. PMID 28434648
- [Background] Balar AV, Galsky MD, Rosenberg JE, Powles T, Petrylak DP, Bellmunt J, Loriot Y, Necchi A, Hoffman-Censits J, Perez-Gracia JL, Dawson NA, van der Heijden MS, Dreicer R, Srinivas S, Retz MM, Joseph RW, Drakaki A, Vaishampayan UN, Sridhar SS, Quinn DI, Duran I, Shaffer DR, Eigl BJ, Grivas PD, Yu EY, Li S, Kadel EE 3rd, Boyd Z, Bourgon R, Hegde PS, Mariathasan S, Thastrom A, Abidoye OO, Fine GD, Bajorin DF; IMvigor210 Study Group. Atezolizumab as first-line treatment in cisplatin-ineligible patients with locally advanced and metastatic urothelial carcinoma: a single-arm, multicentre, phase 2 trial. Lancet. 2017 Jan 7;389(10064):67-76. doi: 10.1016/S0140-6736(16)32455-2. Epub 2016 Dec 8. PMID 27939400
- [Background] Schachter J, Ribas A, Long GV, Arance A, Grob JJ, Mortier L, Daud A, Carlino MS, McNeil C, Lotem M, Larkin J, Lorigan P, Neyns B, Blank C, Petrella TM, Hamid O, Zhou H, Ebbinghaus S, Ibrahim N, Robert C. Pembrolizumab versus ipilimumab for advanced melanoma: final overall survival results of a multicentre, randomised, open-label phase 3 study (KEYNOTE-006). Lancet. 2017 Oct 21;390(10105):1853-1862. doi: 10.1016/S0140-6736(17)31601-X. Epub 2017 Aug 16. PMID 28822576